CLINICAL TRIAL: NCT06335862
Title: Primary pOsterioR TRacheopexy Prevents Collapse of the Trachea in Newborns With Oesophageal AtresIa and Tracheomalacia
Brief Title: Primary Posterior Tracheopexy Prevents Tracheal Collapse
Acronym: PORTRAIT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Erasmus Medical Center (Other); Karolinska University Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); For Wis(h)dom Foundation (funding) (Unknown)
Responsible Party: Principal Investigator, Maud Lindeboom, Principal investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL.84862.041.23
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Oesophageal Atresia With Tracheo-Oesophageal Fistula; Tracheomalacia; Oesophageal Atresia
Keywords: Oesophageal atresia; Tracheomalacia; Primary Posterior Tracheopexy; Respiratory Morbidity
MeSH Terms: conditions — Esophageal atresia with or without tracheoesophageal fistula; Tracheomalacia; Esophageal Atresia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 into either the intervention group (PPT-group) or the wait-and-see group (no-PPT). Since the sutures of the PPT remain in place (in the PPT-group), the participants are allocated to one arm for the duration of the study. After the PPT was or was not performed, the participants will follow the same follow-up schedule.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants, parents/caregivers, investigators and treating healthcare personnel, except for the surgical team performing the OA correction, will be blinded to which study arm the participant is assigned. None of the data gathered is affected by the unblinded surgical team since the primary and key secondary outcome measures are evaluated based on pseudonymised video footage. Furthermore, this video footage is assessed by otolaryngologists who are blinded to the patient and study arm. Moreover, the follow-up and documentation of the secondary endpoints are typically performed by the paediatrician and speech- and language therapists (not the paediatric surgeon or otolaryngologist).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPT-group (Other): Participants allocated to this study arm will undergo the primary posterior tracheopexy (PPT). This PPT is performed concurrently with the primary OA correction. Afterwards, all patients follow the (same) routine follow-up schedule. This treatment is currently used in some centres.
  Interventions: Other: Randomisation between the PPT- and no-PPT-group; Procedure: Primary Posterior Tracheopexy; Diagnostic Test: Preoperative tracheobronchoscopy; Diagnostic Test: Intraoperative tracheobronchoscopy; Diagnostic Test: Postoperative tracheobronchoscopy through the endotracheal tube during extubation; Diagnostic Test: Postoperative tracheobronchoscopy after 2-6 months
- No-PPT-group (Other): Participants allocated to this study arm will undergo the the primary OA correction, without a PPT. Afterwards, all patients follow the (same) routine follow-up schedule. This treatment is also used in some centres.
  Interventions: Other: Randomisation between the PPT- and no-PPT-group; Diagnostic Test: Preoperative tracheobronchoscopy; Diagnostic Test: Intraoperative tracheobronchoscopy; Diagnostic Test: Postoperative tracheobronchoscopy through the endotracheal tube during extubation; Diagnostic Test: Postoperative tracheobronchoscopy after 2-6 months

INTERVENTIONS:
Other: Randomisation between the PPT- and no-PPT-group — Randomisation is performed between two possible treatment options for tracheomalacia in OA patients; the PPT or the wait-and-see policy (no-PPT).
Procedure: Primary Posterior Tracheopexy — The PPT involves fixating the posterior membrane of the trachea to the spinal ligament with sutures, to prevent the trachea from collapsing.
  Arms: PPT-group
Diagnostic Test: Preoperative tracheobronchoscopy — Prior to OA correction, a flexible and a rigid tracheobronchoscopy will be performed, in addition to a flexible tracheobronchoscopy through the endotracheal tube. Preoperative evaluation of TM through a tracheobronchoscopy is part of standard care for all participating centres.
Diagnostic Test: Intraoperative tracheobronchoscopy — After the PPT is performed, or in case of the no-PPT group at the stage of the surgery when the PPT would usually be performed, a flexible tracheobronchoscopy through the endotracheal tube is carried out. This tracheobronchoscopy is routine care for all patients undergoing a PPT, and is additional for patients in the no-PPT-group.
Diagnostic Test: Postoperative tracheobronchoscopy through the endotracheal tube during extubation — A postoperative flexible tracheobronchoscopy is performed in the neonatal or pediatric intensive care unit (ICU), through the endotracheal tube during extubation. This procedure is a study intervention.
Diagnostic Test: Postoperative tracheobronchoscopy after 2-6 months — Two to six months after OA correction, a follow-up flexible and a rigid tracheobronchoscopy will be performed, under general anesthesia in the surgical theatre. This postoperative evaluation of TM through a tracheobronchoscopy is part of standard care for the Karolinska University Hospital and Great Ormond Street Hospital. At the University Medical Centre Utrecht and Erasmus Medical Centre Rotterdam, this tracheobronchoscopy is performed on indication in approximately half of patients. For the other half of patients, this is a study intervention.

SUMMARY:
Introduction: Children born with a blind-ending gullet (oesophagus), or Oesophageal Atresia (OA), need to undergo surgical correction in the first week of life. OA is often accompanied by a weakened windpipe (trachea), known as tracheomalacia (TM). TM entails that the windpipe collapses during expiration. Severe TM can cause respiratory symptoms, including frequent respiratory tract infections and blue spells, that can potentially lead to life-threatening events. In some patients, major secondary surgical treatment may be indicated. This surgical procedure involves widening the trachea (using sutures) to prevent collapse, known as secondary posterior tracheopexy (SPT). Prior to performing this SPT, complications and negative consequences of TM may have already occurred. This may be prevented by performing this procedure during the primary OA correction, called a primary posterior tracheopexy (PPT). The aim of this trial is to determine if a PPT can decrease - or prevent - tracheal collapse in newborns with OA and TM, compared to a wait-and-see policy (no-PPT).

Methods: This is an international multicentre double-blind randomised controlled trial. Seventy eight children with OA type C will be included. Patients will be included after written parental informed consent. Half of the patients will be randomly allocated to the PPT-group and half to the no-PPT-group. The degree and location of TM are evaluated through preoperative, intraoperative and two postoperative videoscopic examinations of the trachea (tracheobronchoscopy). Whether TM symptoms occur is assessed during three routine follow-up consultations until the age of 6 months. The primary outcome is the degree of collapse of the tracheal wall during the intraoperative tracheobronchoscopy (after performing the PPT/no-PPT), measured in percentages.

Risks and burden: Since OA correction with PPT (more recently implemented in centres of expertise) and without PPT (wait-and-see policy) are both accepted and safe treatment options, participating in the trial does not pose an increased risk or burden with regards to the treatment. Performing tracheobronchoscopies may pose a potential burden. However, a tracheobronchoscopy is a routine diagnostic procedure commonly used to safely assess the trachea. Complications of a tracheobronchoscopy are rare. Also, many of the tracheobronchoscopies are routinely performed as part of standard care for these patients, regardless of the trial.

DETAILED DESCRIPTION:
Rationale:

A congenital blind-ending gullet (oesophagus), or Oesophageal Atresia (OA), is very often accompanied by a weakened windpipe (trachea). This is known as tracheomalacia (TM) and entails that the windpipe collapses during expiration. Severe TM can cause increased respiratory morbidity, including frequent respiratory tract infections and blue spells, that can potentially progress to respiratory arrest. Respiratory morbidity poses a significant burden on OA patients, both in the short term and over the course of long-term follow-up. When severe TM is identified, surgical intervention may be necessary. This surgical procedure involves widening the trachea (using sutures) to prevent its collapse, known as a posterior tracheopexy (PT). Prior to performing this secondary PT (SPT), complications and sequelae of TM may have already manifested. Additionally, performing this PT as a secondary operation after the OA correction is a complex surgical procedure in newborns, and poses a significant risk of damaging the recently performed OA anastomosis. This separate, SPT requires several hours of surgery, due to the presence of extensive adhesions. As a result, there has been a growing trend to carry out the PT concurrently with the initial correction of OA, known as a primary posterior tracheopexy (PPT). Previous studies have shown a decrease in respiratory tract infections (RTI's) and brief respiratory unexplained events (BRUE's) following the implementation of a PPT, when compared to patients who did not undergo PPT. However, it is important to note that these studies were predominantly conducted at a single medical center and relied mostly on retrospective data analysis. To address several sources of bias, such as center-specific factors, selection-bias and information bias, a double-blind randomized controlled trial should be conducted.

To accurately evaluate the effects of PPT versus no-PPT (i.e. the percentage of tracheal wall collapse) a tracheobronchoscopy needs to be performed, as it is the only objective measure for this purpose. Tracheobronchoscopy allows for a direct visual examination of the trachea, with a minimal effect on normal airway dynamics, ensuring a reliable evaluation of the impact of the PPT on the tracheal diameter.

Objective: The aim of this trial is to evaluate if a PPT can significantly decrease - or possibly prevent - the collapse of the trachea in newborns with OA and TM, compared to a wait-and-see policy (no-PPT). Additionally, the trial aims to determine whether the observed effect of PPT on tracheal stability is sustained over time.

Design and methodology:

Study design: a double-blind randomised controlled trial. Study population: neonates with oesophageal atresia (OA) and a distal trachea-oesophageal fistula (TOF), with tracheomalacia (TM).

Intervention: randomisation between performing a PPT or no-PPT Randomization, blinding and treatment allocation: Seventy eight patients will be included in this trial. Half of the patients will be randomised into the PPT-group and half into the no-PPT-group. We expect that the number of included patients will be approximately equally distributed among the four participating centres. However, the number of included patients per center is dependent on the number of patients treated by each center during the trial.

All participants, parents/caregivers, investigators and treating healthcare personnel, except for the surgical team performing the OA correction, will be blinded to which trial arm the participant is assigned.

Patient timeline:

* When a child with OA is born, the principal investigator (PI) of the trial is notified.
* Parents/caretakers will be contacted by the researcher/PI. An informed consent meeting is planned with the parents/caretakers, to explain the trial and to discuss possible outcomes or complications.
* If informed consent is obtained, the inclusion and exclusion criteria are checked, based on the observations during a preoperative tracheobronchoscopy (if the patient has TM or not). If the patient is included, randomization will take place in the surgical theatre.
* Based on the outcome of the randomisation, the PPT is either performed, or the PPT is not performed.
* Subsequently, the OA correction is carried out.
* During postoperative extubation (within one week after surgery) the first postoperative tracheobronchoscopy is performed, during extubation, through the endotracheal tube, in the neonatal or paediatric intensive care unit (ICU).
* After 2-6 months, the second postoperative tracheobronchoscopy is be performed under general anaesthesia in the surgical theatre.
* Patients will be followed-up at the outpatient clinic at around 2-3 weeks of age, 3 months of age, and at 6 months of age. This is according to the routine follow-up schedule.

We expect a duration of the inclusion period of 2,5 years. Patients will be included in the trial from the surgery until the 6 month follow-up timepoint. The trial is thus expected to be finished within three years. It will take approximately 6 months after the last inclusion to analyse results and write a scientific report of the (most important) findings.

No interim analysis is planned for efficacy or futility. Nevertheless, a Data Safety Monitoring Board will monitor the safety during the trial.

Burden and risks, benefit and group relatedness:

Burden: To determine whether the PPT is superior in preventing or reducing tracheal collapse, and subsequently respiratory morbidity, compared to no-PPT, a randomized double-blind trial is necessary.

This trial will eliminate dependence on other factors specific to individual centres and provide generalisable results. Importantly, since OA correction with PPT (more recently implemented in centres of expertise) and without PPT (wait-and-see policy) are both accepted and safe treatment options, participating in the trial does not pose an increased risk or burden for the participants with regards to the treatment. However, randomization of patients in this trial can be burdensome as it involves assigning them to either the PPT or no-PPT group based on chance. Parents/caretakers may have preferences or expectations regarding treatment, and being randomized to a specific group may not align with those preferences.

Performing intra- and postoperative tracheobronchoscopies may pose a potential burden during the trial. However, a tracheobronchoscopy is a routine diagnostic procedure commonly used to safely assess the condition of the trachea, even in newborns. Complications arising from a tracheobronchoscopy are rare. An intraoperative tracheobronchoscopy through the ventilation tube is always performed in patients with a PPT as routine care. In patients with ventilatory problems, even without PPT, an intraoperative tracheobronchoscopy can also be routinely performed. In this double-blind randomised trial, all patients will undergo the intra-operative flexible tracheobronchoscopy through the ventilation tube. However, considering the controlled circumstances, there is negligible burden and negligible risk.

After the correction of OA, newborns are typically extubated in the neonatal or paediatric ICU within a few days. During this extubation process, the first postoperative tracheobronchoscopy is conducted through the ventilation tube by a paediatric otorhinolaryngologist, with the presence of the ICU specialist and ICU nurse. Therefore, the burden and risk associated with the tracheobronchoscopy procedure are considered negligible, given the controlled and supervised environment. The second postoperative tracheobronchoscopy may present a burden due to the need for readmission and administration of general anaesthesia in the surgical theatre. However, a routine tracheobronchoscopy in the surgical theatre is often performed in all (Karolinska University Hospital and Great Ormond Street Hospital) or half (University Medical Centre Utrecht and Erasmus Medical Centre Rotterdam) of the OA patients. Thus, only in a small percentage of the trial participants, an extra tracheobronchoscopy is needed. Since the majority of these latter patients undergo an oesophagogastroscopy under general anaesthesia for clinical reasons (e.g. dilatation/eosinophilic oesophagitis), the second postoperative tracheobronchoscopy will be performed during this planned oesophagogastroscopy if possible. The general anaesthesia is administered to safely and effectively perform the tracheobronchoscopy in a controlled and supervised environment. The tracheobronchoscopy is the only objective measure to evaluate the degree of collapse in these patients. This second postoperative tracheobronchoscopy will determine if the observed effect of the PPT on tracheal stability is sustained beyond the first 2 months. Also, this burden is justifiable due to the potential deterioration of tracheal collapse that can occur in the first months following the initial OA correction. Conducting a second postoperative tracheobronchoscopy allows for the identification of these patients. The ability to identify such patients may outweigh the associated risks or added burden of the additional procedure in a small percentage of the trial participants. Moreover, if there is no difference between the intra-operative tracheobronchoscopy and the first and second tracheobronchoscopies, this could mean that in the future, we could sustain with only the (less burdensome) intra- (or first post-) operative tracheobronchoscopy. The respiratory complaints will be evaluated to research if the degree of TM corresponds with the severity of the symptoms.

Group relatedness: The advantage of conducting the primary posterior tracheopexy (PPT) earlier in the treatment process will become evident through the results of this randomised controlled trial (RCT). If the PPT demonstrates superior outcomes, it could lead to a reduction in postoperative complications and interventions, including tracheobronchoscopies under general anaesthesia and additional surgeries for SPT. Conversely, if the SPT yields better results, it could mean fewer patients undergoing unnecessary PPT procedures. The trial will provide valuable insights to guide the optimal timing and approach for tracheopexy in improving patient outcomes/symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of OA with a distal TOF
* Tracheomalacia
* Written informed consent by both parents or legal representatives

Exclusion Criteria:

* Patients with OA without a distal TOF
* Premature neonates <34 weeks
* Endotracheal tube size < 3.0
* Cormack score 3 or 4 as scored by either the otolaryngologist, anesthesiologist, or neonatal/pediatric intensive care specialist
* Patients with a cyanotic cor vitium

Min Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in degree of TM between the PPT-group and no-PPT-group during intraoperative tracheobronchoscopy | Measured by an intraoperative tracheobronchoscopy performed after freeing the trachea and oesophagus (and the PPT) but before the surgical correction of OA, through the ventilation tube
  The difference in the degree of tracheal collapse between the PPT and the no-PPT group measured in percentage of the tracheal diameter

SECONDARY OUTCOMES:
Key secondary outcome: Difference in degree of TM between the PPT-group and no-PPT-group during postoperative tracheobronchoscopy | Measured by a tracheobronchoscopy performed during extubation (approximately 1 day after surgery) and by a tracheobronchoscopy 2-6 months after surgery.
  The difference in the degree of collapse of the tracheal wall between the PPT and the no-PPT group measured in percentages, during:
  * the postoperative flexible tracheobronchoscopy through the ventilation tube during routine extubation in the pediatric or neonatal ICU after approximately 1-3 days,
  * the mostly routine* 2nd postoperative flexible and rigid tracheobronchoscopy that is conducted under general anesthesia in the surgical theatre after approximately 2-6 months. This tracheobronchoscopy serves as a key secondary endpoint and aims to determine whether the effect of PPT is sustained and/or if the TM deteriorates beyond the first 2 months.
    * routinely performed in all patients in Stockholm and London and almost 50% of patients in Utrecht and Rotterdam (the rest of the patients in Utrecht and Rotterdam will undergo this 2nd postoperative tracheobronchoscopy during their routine oesophagogastroscopy (35%) or separately)
Difference in symptoms between the PPT-group and no-PPT-group | During follow-up, starting at the first follow-up consultation at 2-3 months, until the last follow-up consultation at 6 months.
  To investigate the difference between the PPT group and no-PPT group the following endpoints are used:
  The number of respiratory symptoms, the number of RTI's and BRUE's, the number of postoperative complications, the number of hospital admissions and the number of additional conventional, medicinal or surgical interventions, the ventilation duration, and the length of hospital stay in the first six months of life.
Degree of preoperative TM compared to postoperative TM | Comparison between the measurements during the preoperative tracheobronchoscopy and the postoperative tracheobronchoscopy at 2-6 months postoperative.
  The preoperative degree of TM (tracheal wall collapse in percentages) compared to the outcomes of the primary and key secondary endpoints (the intra- and postoperative degree (tracheal wall collapse in percentages) of TM during flexible tracheobronchoscopy through the ventilation tube during extubation in the pediatric or neonatal ICU, and the postoperative tracheobronchoscopy after 2-6 months in the surgical theatre).

CONTACTS AND LOCATIONS:
Overall Officials: John Vlot, MD, PhD, Principal Investigator — Erasmus Medical Center; Jan F Svensson, MD, PhD, Principal Investigator — Karolinska University Hospital; Colin Butler, MD, PhD, Principal Investigator — Great Ormond Street Hospital
Locations (3):
- Netherlands (2):
  - Erasmus Medical Center Rotterdam, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Investigators will strive for publication of results in a peer-reviewed, scientific journal, unreservedly.

REFERENCES:
- [Background] GROSS RE. Atresia of the esophagus. Am J Dis Child (1911). 1947 Sep;74(3):369. No abstract available. PMID 20267729
- [Background] Pedersen RN, Calzolari E, Husby S, Garne E; EUROCAT Working group. Oesophageal atresia: prevalence, prenatal diagnosis and associated anomalies in 23 European regions. Arch Dis Child. 2012 Mar;97(3):227-32. doi: 10.1136/archdischild-2011-300597. Epub 2012 Jan 13. PMID 22247246
- [Background] Macchini F, Parente G, Morandi A, Farris G, Gentilino V, Leva E. Classification of Esophageal Strictures following Esophageal Atresia Repair. Eur J Pediatr Surg. 2018 Jun;28(3):243-249. doi: 10.1055/s-0037-1598656. Epub 2017 Mar 6. PMID 28264202
- [Background] Dodge-Khatami A, Deanovic D, Sacher P, Weiss M, Gerber AC. Clinically relevant tracheomalacia after repair of esophageal atresia: the role of minimal intra-operative dissection and timing for aortopexy. Thorac Cardiovasc Surg. 2006 Apr;54(3):178-81. doi: 10.1055/s-2005-872954. PMID 16639679
- [Background] Kovesi T, Rubin S. Long-term complications of congenital esophageal atresia and/or tracheoesophageal fistula. Chest. 2004 Sep;126(3):915-25. doi: 10.1378/chest.126.3.915. PMID 15364774
- [Background] Sistonen SJ, Pakarinen MP, Rintala RJ. Long-term results of esophageal atresia: Helsinki experience and review of literature. Pediatr Surg Int. 2011 Nov;27(11):1141-9. doi: 10.1007/s00383-011-2980-7. Epub 2011 Sep 30. PMID 21960312
- [Background] Hysinger EB, Panitch HB. Paediatric Tracheomalacia. Paediatr Respir Rev. 2016 Jan;17:9-15. doi: 10.1016/j.prrv.2015.03.002. Epub 2015 Mar 17. PMID 25962857
- [Background] Chetcuti P, Phelan PD. Respiratory morbidity after repair of oesophageal atresia and tracheo-oesophageal fistula. Arch Dis Child. 1993 Feb;68(2):167-70. doi: 10.1136/adc.68.2.167. PMID 8481036
- [Background] Thakkar H, Upadhyaya M, Yardley IE. Bronchoscopy as a screening tool for symptomatic tracheomalacia in oesophageal atresia. J Pediatr Surg. 2018 Feb;53(2):227-229. doi: 10.1016/j.jpedsurg.2017.11.003. Epub 2017 Nov 11. PMID 29217321
- [Background] Koumbourlis AC, Belessis Y, Cataletto M, Cutrera R, DeBoer E, Kazachkov M, Laberge S, Popler J, Porcaro F, Kovesi T. Care recommendations for the respiratory complications of esophageal atresia-tracheoesophageal fistula. Pediatr Pulmonol. 2020 Oct;55(10):2713-2729. doi: 10.1002/ppul.24982. Epub 2020 Aug 7. PMID 32716120
- [Background] Sumida W, Yasui A, Shirota C, Makita S, Okamoto M, Ogata S, Takimoto A, Takada S, Nakagawa Y, Kato D, Gohda Y, Amano H, Guo Y, Hinoki A, Uchida H. Update on aortopexy and posterior tracheopexy for tracheomalacia in patients with esophageal atresia. Surg Today. 2024 Mar;54(3):211-219. doi: 10.1007/s00595-023-02652-6. Epub 2023 Feb 2. PMID 36729255
- [Background] Shieh HF, Smithers CJ, Hamilton TE, Zurakowski D, Rhein LM, Manfredi MA, Baird CW, Jennings RW. Posterior tracheopexy for severe tracheomalacia. J Pediatr Surg. 2017 Jun;52(6):951-955. doi: 10.1016/j.jpedsurg.2017.03.018. Epub 2017 Mar 18. PMID 28385426
- [Background] Shieh HF, Smithers CJ, Hamilton TE, Zurakowski D, Visner GA, Manfredi MA, Baird CW, Jennings RW. Posterior Tracheopexy for Severe Tracheomalacia Associated with Esophageal Atresia (EA): Primary Treatment at the Time of Initial EA Repair versus Secondary Treatment. Front Surg. 2018 Jan 15;4:80. doi: 10.3389/fsurg.2017.00080. eCollection 2017. PMID 29379786
- [Background] van Tuyll van Serooskerken ES, Tytgat SHAJ, Verweij JW, Bittermann AJN, Coenraad S, Arets HGM, van der Zee DC, Lindeboom MYA. Primary Posterior Tracheopexy in Esophageal Atresia Decreases Respiratory Tract Infections. Front Pediatr. 2021 Sep 9;9:720618. doi: 10.3389/fped.2021.720618. eCollection 2021. PMID 34568240
- [Background] Yasui A, Hinoki A, Amano H, Shirota C, Tainaka T, Sumida W, Yokota K, Makita S, Okamoto M, Takimoto A, Nakagawa Y, Uchida H. Thoracoscopic posterior tracheopexy during primary esophageal atresia repair ameliorate tracheomalacia in neonates: a single-center retrospective comparative cohort study. BMC Surg. 2022 Jul 25;22(1):285. doi: 10.1186/s12893-022-01738-1. PMID 35879691
- [Background] Tytgat SHAJ, van Herwaarden-Lindeboom MYA, van Tuyll van Serooskerken ES, van der Zee DC. Thoracoscopic posterior tracheopexy during primary esophageal atresia repair: a new approach to prevent tracheomalacia complications. J Pediatr Surg. 2018 Jul;53(7):1420-1423. doi: 10.1016/j.jpedsurg.2018.04.024. Epub 2018 Apr 27. PMID 29804792
- [Background] Tugcu GD, Soyer T, Polat SE, Hizal M, Emiralioglu N, Yalcin E, Dogru D, Kiper N, Ozcelik U. Evaluation of pulmonary complications and affecting factors in children for repaired esophageal atresia and tracheoesophageal fistula. Respir Med. 2021 May;181:106376. doi: 10.1016/j.rmed.2021.106376. Epub 2021 Mar 28. PMID 33813207
- [Background] Donn SM, Sinha SK. Pulmonary diagnostics. Semin Fetal Neonatal Med. 2017 Aug;22(4):200-205. doi: 10.1016/j.siny.2017.03.006. Epub 2017 Apr 4. PMID 28389088
- [Background] Krishnan U, Mousa H, Dall'Oglio L, Homaira N, Rosen R, Faure C, Gottrand F. ESPGHAN-NASPGHAN Guidelines for the Evaluation and Treatment of Gastrointestinal and Nutritional Complications in Children With Esophageal Atresia-Tracheoesophageal Fistula. J Pediatr Gastroenterol Nutr. 2016 Nov;63(5):550-570. doi: 10.1097/MPG.0000000000001401. PMID 27579697
- [Derived] van Stigt MJB, van Hal ARL, Bittermann AJN, Butler CR, Ceelie I, Cianci D, de Coppi P, Gahm C, Hut JE, Joosten KFM, Lemmers PMA, Mullassery D, Nandi R, Pullens B, Staals LM, Svensson JF, Tytgat SHAJ, van de Ven PM, Wijnen RMH, Vlot J, Lindeboom MYA. Does primary posterior tracheopexy prevent collapse of the trachea in newborns with oesophageal atresia and tracheomalacia? A study protocol for an international, multicentre randomised controlled trial (PORTRAIT trial). BMJ Open. 2024 Dec 12;14(12):e087272. doi: 10.1136/bmjopen-2024-087272. PMID 39672574